CLINICAL TRIAL: NCT06647589
Title: Efficacy of Acceptance and Commitment Therapy on Religiously Oriented Obsessive-Compulsive Disorder
Brief Title: Acceptance and Commitment Therapy for Religious OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Johnson, Graduate Student, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300013565-001; UAB (Other: UAB)
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-03

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: scrupulosity; religion; acceptance and commitment therapy; obsessive-compulsive disorder; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and Commitment Therapy (Experimental): Participants will receive twelve consecutive weeks of acceptance and commitment therapy
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — participants will then receive ACT-based individual therapy weekly for twelve weeks.

SUMMARY:
The purpose of the study is to examine the effects and feasibility of a specific form of psychotherapy, acceptance and commitment therapy (ACT), on religiously oriented obsessive and compulsive disorder (OCD).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Meet cutoff scores for scrupulosity

Exclusion Criteria:

* Presence of psychotic symptoms within six months of screening
* Current suicidal/homicidal plan/intent and/or a suicide/homicide attempt within 6 months of screening
* Non-suicidal self-injury within 6 months of screening
* Narcotics use within 3 months of screening
* Purging/restricting behavior within 3 months of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Scrupulosity Obsessions and Compulsions Scale | At baseline, 4 weeks, 8 weeks, and post-intervention (12 weeks)
  The Scrupulosity Obsessions and Compulsions Scale (SOCS) is a 10-item scale that asks participants how often they experience religious OCD obsessions and compulsions. The questions are asked on a scale ranging from 0 (Very Rarely) to 5 (Very Often).
Experiential Avoidance Rating Scale | At baseline, 4 weeks, 8 weeks, and post-intervention (12 weeks)
  The Experiential Avoidance Rating Scale (EARS) is a 6-item scale that asks participants how true statements about avoiding experiences are for them. The questions are asked on a scale ranging from 1 (Never True) to 5 (Very Often True).

SECONDARY OUTCOMES:
Centrality of Religiosity Scale - Interreligious 20 | Pre and post intervention which in general lasts 12 weeks
  The Centrality of Religiosity Scale - Interreligious 20 (CRSi-20) is a 20-item scale assessing religiosity across 5 dimensions (Intellect, Ideology, Public practice, Private practice, Experience). The questions are asked on scales ranging from Never to Several times a day, Never to Very often, and Not at all to Very much so.
Yale-Brown Obsessive and Compulsive Scale - Self Report | Pre and post intervention which in general lasts 12 weeks
  The Yale-Brown Obsessive and Compulsive Scale (Y-BOCS) is a 12-item scale that asks participants whether they experience various OCD obsessions and compulsions. Participants are then asked how much time is spent on these obsessions and compulsions, whether they give in to the urge to perform compulsions, how strong the drive is to give in to compulsions, how they would feel if they were prevented from engaging in compulsions, and how much the compulsions and avoidance of compulsions interfere with their functioning.
Patient Health Questionnaire - 9 | Pre and post intervention which in general lasts 12 weeks
  The Patient Health Questionnaire (PHQ-9) is a 9-item scale that asks participants how often they have been bothered by aspects of depressive symptoms. The questions are asked on a scale ranging from 0 (Not at all) to 5 (Nearly every day).
Generalized Anxiety Disorder - 7 | Pre and post intervention which in general lasts 12 weeks
  The Generalized Anxiety Disorder Scale (GAD-7) is a 7-item scale that asks participants how often they have been bothered by statements capturing aspects of anxiety. The questions are asked on a scale ranging from 0 (Not at all) to 3 (Nearly every day).
The Intrinsic Spirituality Scale | Pre and post intervention which in general lasts 12 weeks
  The Intrinsic Spirituality Scale is a 6-item scale that asks participants about aspects of their spirituality.
Psy-Flex | Pre and post intervention which in general lasts 12 weeks
  The Psyflex questionnaire is a 6-item scale that measures aspects of psychological flexibility. The questions are asked on a scale ranging from very seldom to often.
Almost Perfect Scale - Revised | Pre and post intervention which in general lasts 12 weeks
  The Almost Perfect Scale - Revised is a 23-item scale that asks participants their agreement on items capturing perfectionism. The questions are asked on a scale ranging from 1 (Strongly disagree) to 7 (Strongly agree).
The Alcohol Use Disorders Identification Test | Pre and post intervention which in general lasts 12 weeks
  The Alcohol Use Disorders Identification Test (AUDIT) is a 10-item scale that asks participants about their alcohol consumption.
National Institute on Drug Abuse Screener | Pre and post intervention which in general lasts 12 weeks
  National Institute on Drug Abuse Screener (NIDA) is a 1-item scale that asks participants how often they use a variety of substances. The questions are asked on a scale ranging from Never to Daily or Almost Daily.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes